CLINICAL TRIAL: NCT01620398
Title: The Brazilian Cardioprotective Nutritional Program to Reduce Events and Risk Factors in Secondary Prevention for Cardiovascular Disease
Brief Title: Brazilian Cardioprotective Nutritional Program Trial
Acronym: BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCDT
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular diseases; secondary prevention; diet
MeSH Terms: conditions — Cardiovascular Diseases | interventions — 4-azidobenzylcarazolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BALANCE group (Experimental): BALANCE Program is composed by 3 concepts: a) a diet composed of 50-60% of energy from carbohydrate, 10-15% of energy from protein; 25-35% of energy from fat (<7% saturated fatty acid; <10% polyunsaturated fatty acid; <20% monounsaturated fatty acid, <1% trans fatty acid), <200 mg/day of cholesterol, 20-30 g/day of fiber and <2400 mg/day of sodium; b) Nutrition education program based on ludic strategies and indication of affordable foods; c) An intense follow up by individual and group visits and phone calls.
  Interventions: Behavioral: BALANCE
- Control Diet group (Active Comparator): generalized advices to follow a low fat, low energy, low sodium and low cholesterol diet are given.
  Interventions: Behavioral: Control diet

INTERVENTIONS:
Behavioral: BALANCE
  Other Names: DICA Br;; PABC;
  Arms: BALANCE group
Behavioral: Control diet — Participants will be encourage to follow a generalized diet counseling prepared by dietitians based on low fat, low energy, low sodium and low cholesterol diets. They will receive a common folder composed by lists of foods that should be preferred or avoided. For example, avoidance of ultra processed foods, preference for boiled and baked foods rather than fried foods and recommendation of having at least five meals a day. This folder is equivalent of several that are given on ambulatories or hospital of Brazilian public health.
  Arms: Control Diet group

SUMMARY:
There are no studies exploring the benefits of a diet composed of typical Brazilian food in the secondary prevention of cardiovascular diseases. Randomized studies show that the Mediterranean diet is beneficial for patients with established cardiovascular disease or in risk for CVD development. Indeed, nutritional composition of the Mediterranean Diet is one of main references for dietary guidelines for treatment and prevention of CVD in Brazil and the world. However, in many countries, such as Brazil, most foods of the Mediterranean diet are not widely available, may be expensive or are not part of population eating habits. So, the prescription of the Mediterranean diet intervention for cardiovascular disease to the Brazilian population may not be feasible, leading to a low adherence. In this context, patients with established CVD have a low compliance to nutritional prescription. The BALANCE Program, considers 3 concepts: a) A dietary prescription guided by nutritional content recommendations from the Brazilian national guidelines; b) A nutritional education program based on fun, playful strategies and suggestions of affordable foods; and c) Intensive follow-up through one-on-one visits, group sessions, and phone calls. This is the first proposal to use these concepts concurrently with the objective to increase adherence of secondary prevention patients to the diet proposed by the guidelines. Therefore, The primary outcome is a composite of death (any cause), cardiac arrest, acute myocardial infarction, stroke, myocardial revascularization, amputation for peripheral arterial disease, or hospitalization for unstable angina.

DETAILED DESCRIPTION:
The BALANCE Program will investigate the effect of the Program in reducing cardiovascular events, such as cardiac arrest, acute myocardial infarction, stroke, myocardial revascularization, amputation for peripheral arterial disease, hospitalization for unstable angina, or death in patients with established cardiovascular disease. Moreover the aim is to evaluate the effect of the dietary program on reducing cardiovascular risk factors, such as body mass index, waist circumference, blood pressure, total cholesterol, low density lipoprotein (LDL), triglycerides and fasting glucose. Also the objective is to compare the dietary patterns after interventions, the effect of the intervention among nutrients and energy consumption and, finally, to evaluate the BALANCE Program comprehension.

The BALANCE Program is a randomized, multicenter, national trial with allocation concealment and intention-to-treat analysis. The elegibility criteria is patients aged 45 years or more with any evidence of established cardiovascular disease to the BALANCE program or control groups. BALANCE Program is composed by 3 concepts: a) a diet that provides 50-60% of energy from carbohydrate, 10-15% from protein, 25-35% from total fat, <7% from saturated fatty acids, <10% polyunsaturated fatty acids, <20% monounsaturated fatty acids, <1% trans fats, <200 mg/day cholesterol, 20-30 g/day fiber, and <2,400 mg/day sodium; b) Nutrition education program based on ludic strategies and indication of affordable foods; c) An intense follow up by individual and group visits and phone calls. For Control group, generalized advices to follow a low fat, low energy, low sodium and low cholesterol diet are given. The primary composite outcome is the occurrence of of death (any cause), cardiac arrest, acute myocardial infarction, stroke, myocardial revascularization, amputation for peripheral arterial disease or hospitalization for unstable angina. Blinded assessors will adjudicate clinical events and analysis will follow the intention-to-treat principle. Were enrolled 2534 patients in 35 sites. Enrollment was open in March 2013 and ended in March 2015 and patients will be followed up to 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Any evidence of coronary artery disease (CAD) over the preceding 10 years, as defined by any of the following criteria:

  * defined by previous myocardial infarction,
  * stable or unstable angina,
  * history of atherosclerotic stenosis ≥70% of the diameter of any coronary artery on conventional or computed tomographic (CT) coronary angiography,
  * history of angioplasty, stenting, or coronary artery bypass surgery)
* Any evidence of stroke in the preceding 10 years
* Peripheral Arterial Disease over the preceding 10 years, as defined by any of the following criteria:

  * ankle/arm ratio <0.9 of systolic blood pressure in either leg at rest, angiography or Doppler demonstrating >70% stenosis in a cardiac artery,
  * intermittent claudication,
  * vascular surgery for atherosclerotic disease,
  * amputation due to atherosclerotic disease,
  * aortic aneurysm

Exclusion Criteria:

* Refusal to provide Informed Consent Statement
* neurocognitive or psychiatric condition that may hinder collection of reliable clinical data (defined at the trial investigator's discretion)
* Life expectancy less than 6 months
* Pregnancy or lactation
* Liver failure with a history of encephalopathy or anasarca
* Renal Failure with indication for dialysis
* Congestive heart failure
* Previous organ transplantation
* Wheelchair use
* Any restrictions to receiving an oral diet.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2534 (Actual)
Dates: Start 2013-03-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Composity of Major Cardiovascular Events | up to 48 month
  The primary composite outcome will be the occurrence of any of the following cardiovascular events: cardiac arrest, acute myocardial infarction, stroke, myocardial revascularization, amputation for peripheral arterial disease, hospitalization for unstable angina, cardiovascular death, or death from any cause.
  The Clinical Endpoints Committee (CEC) will be responsible for adjudication of primary composite outcome components. All suspected events will be entered into the CEC tracking database and independently reviewed by two CEC physicians. If the two adjudicators agree, event adjudication will be considered complete. If there is disagreement, the final decision will be made by a third, independent adjudicator.
  It will be reported in events per person-years and crude rate per 1000 person-years.

SECONDARY OUTCOMES:
Total cholesterol (mg/dl) | up to 48 month
  For biochemical analyses blood samples will be collected and handled according to routine hospital practice. All participants will be fasted for at least 12 hours before phlebotomy. It will be analyzed over time by repeated-measures analysis of variance using a mixed model or generalized estimating equations.
LDL - cholesterol (mg/dl) | up to 48 month
  For biochemical analyses blood samples will be collected and handled according to routine hospital practice. It will be estinated by Friedewald formula. All participants will be fasted for at least 12 hours before phlebotomy. It will be analyzed over time by repeated-measures analysis of variance using a mixed model or generalized estimating equations
Fasting glucose (mg/dL) | up to 48 month
  For biochemical analyses blood samples will be collected and handled according to routine hospital practice. All participants will be fasted for at least 12 hours before phlebotomy. It will be analyzed over time by repeated-measures analysis of variance using a mixed model or generalized estimating equations.
Blood pressure (mmHg) | up to 48 month
  It will be analyzed over time by repeated-measures analysis of variance using a mixed model or generalized estimating equations
Body-mass index (kg/m2) | up to 48 month
  Compose by body weight (in kilograms) and body height (in meters), reported in kg/m².It will be analyzed over time by repeated-measures analysis of variance using a mixed model or generalized estimating equations.
waist circumference (cm) | up to 48 month
  It will be analyzed over time by repeated-measures analysis of variance using a mixed model or generalized estimating equations. The values of the circumferences will be expressed in centimeters (cm). The waist circumference should be measured through the midpoint between the lower border of the costal arch and the iliac crest in the medial axillary line.
Triglycerides (mg/dL) | up to 48 month
  For biochemical analyses blood samples will be collected and handled according to routine hospital practice. All participants will be fasted for at least 12 hours before phlebotomy.
  It will be analyzed over time by repeated-measures analysis of variance using a mixed model or generalized estimating equations
isolated occurrence of cardiovascular events | up to 48 month
  cardiac arrest, acute myocardial infarction, stroke, myocardial revascularization, amputation for peripheral arterial disease, hospitalization for unstable angina, or isolated cardiovascular death.
  The Clinical Endpoints Committee (CEC) will be responsible for adjudication of primary composite outcome components. All suspected events will be entered into the CEC tracking database and independently reviewed by two CEC physicians. If the two adjudicators agree, event adjudication will be considered complete. If there is disagreement, the final decision will be made by a third, independent adjudicator.
  It will be reported in events per person-years and crude rate per 1000 person-years.
isolated cardiovascular death or death from any cause | up to 48 month
  isolated cardiovascular death or death from any cause The Clinical Endpoints Committee (CEC) will be responsible for adjudication of primary composite outcome components. All suspected events will be entered into the CEC tracking database and independently reviewed by two CEC physicians. If the two adjudicators agree, event adjudication will be considered complete. If there is disagreement, the final decision will be made by a third, independent adjudicator.
  It will be reported in events per person-years and crude rate per 1000 person-years.
nutrient and energy intake analysis | up to 48 month
  It will be analyzed over time by repeated-measures analysis of variance using a mixed model or generalized estimating equations.
  Dietary intake data was assessed from two 24-hour recall from each visit, collected by trained interviewers. Nutrients will be present in grams/day and in % of calories and energy in Kcal.
dietary pattern analysis | up to 48 month
  a posteriori and/or a priori analysis. The dietary intake data will be obtain from two 24-hour recalls and the nutrient variability was adjusted by the Multiple Source Method (MSM). Dietary patterns were obtained by principal component analysis, and the scores were categorized into tertiles.
BALANCE Program comprehension | up to 48 month
  Each telephone monitoring will address questions about the nutritional guidelines received by the patient in order to identify the understanding of the information after the follow-up visit. The answers will be imputed in an electronic system developed for the telephone monitoring of DICA Br.
  It will be analysed by chi-square and/or regression analysis.
Cost-effectiveness analysis of clinical events (U$/events) | up to 36 month
  A cost-effectiveness analysis will be performed taking into consideration the societal perspective. BALANCE diet cost and the healthcare expenditures will be estimated in both intervention and control groups among individuals who were adherent to BALANCE study protocol.
  Clinical outcomes will determine the effectiveness of the BALANCE study. The expected clinical outcomes are death, cardiac arrest, myocardial infarction, stroke, myocardial revascularization, amputation, or angina. Differences between the cost-effectiveness rates fwill determine the cost-effectiveness analysis of clinical events. External validity will be performed using sensibility analyses.
Cost-effectiveness analysis of diet quality (U$/DQIscore) | up to 36 month
  A cost-effectiveness analysis will be performed taking into consideration the societal perspective. BALANCE diet cost and the healthcare expenditures will be estimated in both intervention and control groups among individuals who were adherent to BALANCE study protocol.
  Diet quality will be obtained by diet quality index (DQI) and will determine the effectiveness of the BALANCE study.
  Differences between the cost-effectiveness rates will determine the Cost-effectiveness analysis of diet quality External validity will be performed using sensibility analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardete Berwanger, NC, PhD, Principal Investigator — Hospital do Coração; Otávio Berwanger, MD, PhD, Study Director — Hospital do Coração; Rafael M Soares, NC, MSc, Study Chair — Hospital do Coração; Rosana P Costa, NC, MSc, Study Chair — Hospital do Coração; Maria B Ross-Fernandes, NC, MSc, Study Chair — Hospital do Coração; Enilda S Lara, NC, PhD, Study Chair — Hopsital do Coração; Camila R Torreglosa, NC, MSc, Study Chair — Hospital do Coração; Ângela C Bersch-Ferreira, NC, MSc, Study Chair — Hospital do Coração; Jacqueline T da Silva, NC, Study Chair — Hospital do Coração; Andrea P Galante, NC, PhD, Study Chair — Hospital do Coração
Locations (35):
- Brazil (35):
  - Universidade Federal de Alagoas, Maceió, Alagoas
  - Hospital Universitário Francisca Mendes, Manaus, Amazonas
  - Hospital de Messejana, Fortaleza, Ceará
  - Universidade de Fortaleza, Fortaleza, Ceará
  - Hospital Universitário Professor Edgard Santos / ENUFBA / UFBA, Salvador, Estado de Bahia
  - Hospital das Clínicas de Goiânia, Goiânia, Goiás
  - Hospital Universitário Federal Presidente Dutra, São Luiz, Maranhão
  - Universidade Federal do Mato Grosso, Cuiabá, Mato Grosso
  - Hospital Universitário Maria Aparecida Pedrossian, Campo Grande, Mato Grosso do Sul
  - Universidade Federal de Viçosa, Viçosa, Minas Gerais
  - Hospital de Clínicas da Universidade Federal do Paraná, Curitiba, Paraná
  - Hospital Universitário Alcides Carneiro, Campina Grande, Paraíba
  - Hospital das Clínicas Gaspar Viana, Belém, Pará
  - Pronto Socorro Cardiológico Universitário de Pernambuco, Recife, Pernambuco
  - IECAC, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Ana Bezerra, Santa Cruz, Rio Grande do Norte
  - URCAMP, Bagé, Rio Grande do Sul
  - Hospital Universitário AESC, Canoas, Rio Grande do Sul
  - BIOSERV, Passo Fundo, Rio Grande do Sul
  - Universidade Federal de Pelotas, Pelotas, Rio Grande do Sul
  - COTENUT, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da Pontifícia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Associação Veranense de Assistência em Saúde (AVAES), Veranópolis, Rio Grande do Sul
  - Universidade Vale do Itajaí, Itajaí, Santa Catarina
  - Hospital São Lucas, Aracaju, Sergipe
  - Hospital Universitário FUFSE, Aracaju, Sergipe
  - Universidade Federal de Tocantins, Palmas, Tocantins
  - Hospital Universitário de Brasília, Brasília
  - Hospital Universitario Pedro Ernesto, Rio de Janeiro
  - Instituto Nacional de Cardiologia, Rio de Janeiro
  - Hospital do Coração, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Universidade Federal de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almeida AP, Lopes LJ, Bersch-Ferreira AC, Torreglosa CR, Marcadenti A, Weber B, Bressan J, Hermsdorff HHM. Insulin resistance mediate the association between leucine intake, dietary glycemic index, and type 2 diabetes in secondary cardiovascular prevention: path analysis from Brazilian cardioprotective nutritional (BALANCE) program. Eur J Nutr. 2025 Mar 29;64(3):140. doi: 10.1007/s00394-025-03653-6. PMID 40156624
- [Derived] Bersch-Ferreira AC, Hall WL, Santos RHN, Torreglosa CR, Sampaio G, Tereza da Silva J, Alves R, Ross MB, Gehringer MO, Kovacs C, Marcadenti A, Magnoni D, Weber B, Rogero MM. The effect of the a regional cardioprotective nutritional program on inflammatory biomarkers and metabolic risk factors in secondary prevention for cardiovascular disease, a randomised trial. Clin Nutr. 2021 Jun;40(6):3828-3835. doi: 10.1016/j.clnu.2021.04.035. Epub 2021 Apr 28. PMID 34130029
- [Derived] de Brito Goncalves Nascimento L, Sahade V, Weber B, Pinheiro JMF, Dias LPP, Figueiredo Neto JA, Carlos Sobral Sousa A, Pinho CPS, Luna AB, Vasconcelos SML, Dantas CF, Penafort AM, Carlos DMO, Daltro C. Diabetic Patients with Cardiovascular Disease Show More Metabolic Syndrome than Nondiabetic Patients: Multicentric Study in the Northeast of Brazil. Metab Syndr Relat Disord. 2021 May;19(4):233-239. doi: 10.1089/met.2020.0064. Epub 2021 Feb 1. PMID 33523760
- [Derived] Alves da Silva R, Bersch-Ferreira AC, Gehringer MO, Ross-Fernandes MB, Kovacs do Amaral C, Lin Wang HT, Lima PH, de Lima PA, Franca JI, Weber B, Magnoni CD, Rogero MM. Effect of qualitative and quantitative nutritional plan on gene expression in obese patients in secondary prevention for cardiovascular disease. Clin Nutr ESPEN. 2021 Feb;41:351-359. doi: 10.1016/j.clnesp.2020.11.002. Epub 2020 Nov 26. PMID 33487289
- [Derived] Weber B, Bersch-Ferreira AC, Torreglosa CR, Marcadenti A, Lara ES, da Silva JT, Costa RP, Santos RHN, Berwanger O, Bosquetti R, Pagano R, Mota LGS, de Oliveira JD, Soares RM, Galante AP, da Silva SA, Zampieri FG, Kovacs C, Amparo FC, Moreira P, da Silva RA, Dos Santos KG, Monteiro AS, Paiva CCJ, Magnoni CD, Moreira ASB, Pecanha DO, Missias KCS, de Paula LS, Marotto D, Souza P, Martins PRT, Dos Santos EM, Santos MR, Silva LP, Torres RS, Barbosa SNAA, de Pinho PM, de Araujo SHA, Verissimo AOL, Guterres AS, Cardoso AFR, Palmeira MM, de Ataide BRB, Costa LPS, Marinho HA, de Araujo CBP, Carvalho HMS, Maquine RO, Caiado AC, de Matos CH, Barretta C, Specht CM, Onofrei M, Bertacco RTA, Borges LR, Bertoldi EG, Longo A, Ribas BLP, Dobke F, Pretto ADB, Bachettini NP, Gastaud A, Necchi R, Souza GC, Zuchinali P, Fracasso BM, Bobadra S, Sangali TD, Salamoni J, Garlini LM, Shirmann GS, de Los Santos MLP, Bortonili VMS, Dos Santos CP, Braganca GCM, Ambrozio CL, E Lima SB, Schiavini J, Napparo AS, Boemo JL, Nagano FEZ, Modanese PVG, Cunha NM, Frehner C, da Silva LF, Formentini FS, Ramos MEM, Ramos SS, Lucas MCS, Machado BG, Ruschel KB, Beiersdorf JR, Nunes CE, Rech RL, Damiani M, Berbigier M, Poloni S, Vian I, Russo DS, Rodrigues JA, de Moraes MAP, da Costa LM, Boklis M, El Kik RM, Adorne EF, Teixeira JM, Trescastro EP, Chiesa FL, Telles CT, Pellegrini LA, Reis LF, Cardoso RGM, Closs VE, Feres NH, da Silva NF, Silva NE, Dutra ES, Ito MK, Lima MEP, Carvalho APPF, Taboada MIS, Machado MMA, David MM, Junior DGS, Dourado C, Fagundes VCFO, Uehara RM, Sasso S, Vieira JSO, de Oliveira BAS, Pereira JL, Rodrigues IG, Pinho CPS, Sousa ACS, Almeida AS, de Jesus MT, da Silva GB, Alves LVS, Nascimento VOG, Vieira SA, Coura AGL, Dantas CF, Leda NMFS, Medeiros AL, Andrade ACL, Pinheiro JMF, de Lima LRM, Sabino LS, de Souza CVS, Vasconcelos SML, Costa FA, Ferreira RC, Cardoso IB, Navarro LNP, Ferreira RB, Junior AES, Silva MBG, Almeida KMM, Penafort AM, de Queiros APO, Farias GMN, Carlos DMO, Cordeiro CGNC, Vasconcelos VB, de Araujo EMVMC, Sahade V, Ribeiro CSA, Araujo GA, Goncalves LB, Teixeira CS, Silva LMAJ, da Costa LB, Souza TS, de Jesus SO, Luna AB, da Rocha BRS, Santos MA, Neto JAF, Dias LPP, Cantanhede RCA, Morais JM, Duarte RCL, Barbosa ECB, Barbosa JMA, de Sousa RML, Dos Santos AF, Teixeira AF, Moriguchi EH, Bruscato NM, Kesties J, Vivian L, de Carli W, Shumacher M, Izar MCO, Asoo MT, Kato JT, Martins CM, Machado VA, Bittencourt CRO, de Freitas TT, Sant'Anna VAR, Lopes JD, Fischer SCPM, Pinto SL, Silva KC, Gratao LHA, Holzbach LC, Backes LM, Rodrigues MP, Deucher KLAL, Cantarelli M, Bertoni VM, Rampazzo D, Bressan J, Hermsdorff HHM, Caldas APS, Felicio MB, Honorio CR, da Silva A, Souza SR, Rodrigues PA, de Meneses TMX, Kumbier MCC, Barreto AL, Cavalcanti AB. Implementation of a Brazilian Cardioprotective Nutritional (BALANCE) Program for improvement on quality of diet and secondary prevention of cardiovascular events: A randomized, multicenter trial. Am Heart J. 2019 Sep;215:187-197. doi: 10.1016/j.ahj.2019.06.010. Epub 2019 Jun 21. PMID 31349110
- [Derived] da Silva A, Caldas APS, Hermsdorff HHM, Bersch-Ferreira AC, Torreglosa CR, Weber B, Bressan J. Triglyceride-glucose index is associated with symptomatic coronary artery disease in patients in secondary care. Cardiovasc Diabetol. 2019 Jul 11;18(1):89. doi: 10.1186/s12933-019-0893-2. PMID 31296225
- [Derived] Tereza da Silva J, Bersch-Ferreira AC, Torreglosa CR, Weber B, Levy RB. Development of a dietary index based on the Brazilian Cardioprotective Nutritional Program (BALANCE). Nutr J. 2018 May 4;17(1):49. doi: 10.1186/s12937-018-0359-5. PMID 29728114
- [Derived] Weber B, Bersch-Ferreira AC, Torreglosa CR, Ross-Fernandes MB, da Silva JT, Galante AP, Lara Ede S, Costa RP, Soares RM, Cavalcanti AB, Moriguchi EH, Bruscato NM, Kesties, Vivian L, Schumacher M, de Carli W, Backes LM, Reolao BR, Rodrigues MP, Baldissera DM, Tres GS, Lisboa HR, Bem JB, Reolao JB, Deucher KL, Cantarelli M, Lucion A, Rampazzo D, Bertoni V, Torres RS, Verrissimo AO, Guterres AS, Cardos AF, Coutinho DB, Negrao MG, Alencar MF, Pinho PM, Barbosa SN, Carvalho AP, Taboada MI, Pereira SA, Heyde RV, Nagano FE, Baumgartner R, Resende FP, Tabalipa R, Zanini AC, Machado MJ, Araujo H, Teixeira ML, Souza GC, Zuchinali P, Fracasso BM, Ulliam K, Schumacher M, Pierotto M, Hilario T, Carlos DM, Cordeiro CG, Carvalho DA, Goncalves MS, Vasconcelos VB, Bosquetti R, Pagano R, Romano ML, Jardim CA, de Abreu BN, Marcadenti A, Schmitt AR, Tavares AM, Faria CC, Silva FM, Fink JS, El Kik RM, Prates CF, Vieira CS, Adorne EF, Magedanz EH, Chieza FL, Silva IS, Teixeira JM, Trescastro EP, Pellegrini LA, Pinto JC, Telles CT, Sousa AC, Almeida AS, Costa AA, Carmo JA, Silva JT, Alves LV, Sales SO, Ramos ME, Lucas MC, Damiani M, Cardoso PC, Ramos SS, Dantas CF, Lopes AG, Cabral AM, Lucena AC, Medeiros AL, Terceiro BB, Leda NM, Baia SR, Pinheiro JM, Cassiano AN, Melo AN, Cavalcanti AK, Souza CV, Queiroz DJ, Farias HN, Souza LC, Santos LS, Lima LR, Hoffmann MS, Ribeiro AS, Vasconcelos DF, Dutra ES, Ito MK, Neto JA, Santos AF, Sousa RM, Dias LP, Lima MT, Modanesi VG, Teixeira AF, Estrada LC, Modanesi PV, Gomes AB, Rocha BR, Teti C, David MM, Palacio BM, Junior DG, Faria EH, Oliveira MC, Uehara RM, Sasso S, Moreira AS, Cadinha AC, Pinto CW, Castilhos MP, Costa M, Kovacs C, Magnoni D, Silva Q, Germini MF, da Silva RA, Monteiro AS, dos Santos KG, Moreira P, Amparo FC, Paiva CC, Poloni S, Russo DS, Silveira IV, Moraes MA, Boklis M, Cardoso QI, Moreira AS, Damaceno AM, Santos EM, Dias GM, Pinho CP, Cavalcanti AC, Bezerra AS, Queiroga AV, Rodrigues IG, Leal TV, Sahade V, Amaral DA, Souza DS, Araujo GA, Curvello K, Heine M, Barretto MM, Reis NA, Vasconcelos SM, Vieira DC, Costa FA, Fontes JM, Neto JG, Navarro LN, Ferreira RC, Marinho PM, Abib RT, Longo A, Bertoldi EG, Ferreira LS, Borges LR, Azevedo NA, Martins CM, Kato JT, Izar MC, Asoo MT, de Capitani MD, Machado VA, Fonzar WT, Pinto SL, Silva KC, Gratao LH, Machado SD, de Oliveira SR, Bressan J, Caldas AP, Lima HC, Hermsdorff HH, Saldanha TM, Priore SE, Feres NH, Neves Ade Q, Cheim LM, Silva NF, Reis SR, Penafort AM, de Queiros AP, Farias GM, de los Santos ML, Ambrozio CL, Camejo CN, dos Santos CP, Schirmann GS, Boemo JL, Oliveira RE, Lima SM, Bortolini VM, Matos CH, Barretta C, Specht CM, de Souza SR, Arruda CS, Rodrigues PA, Berwanger O. The Brazilian Cardioprotective Nutritional Program to reduce events and risk factors in secondary prevention for cardiovascular disease: study protocol (The BALANCE Program Trial). Am Heart J. 2016 Jan;171(1):73-81.e1-2. doi: 10.1016/j.ahj.2015.08.010. Epub 2015 Aug 15. PMID 26699603